CLINICAL TRIAL: NCT05773651
Title: Rare Tumours in Children and Adolescents (STEP 2.0) - Register for the Documentation of Rare Tumours in Children and Adolescents
Brief Title: Rare Tumours in Children and Adolescents (STEP)
Acronym: STEP 2 0
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: STEP 2.0
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Rare Diseases
Keywords: Epidemiological data collection; Rare tumors in children; Rare tumors in adolescents; Clinical data collection
MeSH Terms: conditions — Rare Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rare tumor disease: Prospective epidemiological and clinical data collection of subjects with diagnosis of a rare solid tumor.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The data collection includes, among other things: Diagnosis of the rare tumor (pathological findings/ reference pathological findings), full name, birth date, gender, clinical registry inclusion and exclusion criteria met - yes / no, signed declaration of consent-yes / no, if yes: date of signature

SUMMARY:
The aim of the STEP registry is to collect and evaluate experience and data on the diagnosis and treatment of rare childhood tumors in order to use the knowledge gained to improve the treatment prospects for our patients. The rarity of a disease should not be a disadvantage for the young patients.

DETAILED DESCRIPTION:
The objective of the STEP registry is to optimise the diagnosis and treatment of patients with rare tumour diseases in childhood and adolescence. Therefore, a continuous prospective collection of clinical data on rare paediatric tumours is conducted to improve the understanding of these tumours. Beyond analysis of clinical data, further scientific research on the biological and molecular genetic characteristics of these tumours is performed. These data and a close collaboration with international partners, especially the European EXPeRT group, enable the improvement of treatment recommendations for these tumours along with establishment a global interdisciplinary network of rare tumour specialists.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a rare solid tumor
* Age at diagnosis: Neonatal period to 18 years (In the case of young adults, registration in the database and/or referral to advisory contact persons within the framework of the competence network can take place upon request and after declaration of consent.)
* Information, education, written consent of the patient or the guardian
* Not recorded in any of the existing clinical studies/ registers of the German Society for Pediatric Oncology and Hematology (GPOH)

Exclusion Criteria:

* Registration of the tumor diagnosis in a prospective therapy study/ another clinical registry of the GPOH
* Lack of information, explanation and/or written consent of the patient or the legal guardian.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with rare solid tumors from primary care clinic, university hospitals, specialty centers, ...
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2055-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  Period between study entry and failure of induction therapy, recurrence or death from any cause is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Brecht, PD Dr. med., Study Director — University Hospital Tübingen; Dominik Schneider, Prof. Dr. med., Study Director — Clinic for Pediatric and Adolescent Medicine at Dortmund Hospital
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The STEP Register will provide data in a pseudonymised manner to national and international databases set up to optimize the diagnosis and treatment of rare tumors in children and adolescents
Time Frame: Data will become available after analysis and unlimited.

REFERENCES:
- See also: Related Info — http://www.seltene-tumoren.de/